CLINICAL TRIAL: NCT01030939
Title: A Single-blind, Randomised, Placebo-controlled, Parallel Group Study to Investigate Safety, Tolerability, Pharmacokinetics and the Effects on Cardiac Function of Repeat Oral Doses of SB-649868 in Adult and Elderly Healthy Volunteers
Brief Title: Study to Investigate Safety, Tolerability, Pharmacokinetics and Cardiac Function After Repeat Doses of SB-649868 in Healthy-volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112861
Record Dates: First submitted 2009-11-12; First posted 2009-12-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Sleep Disorders
Keywords: Healthy volunteers; Men and women; adults and elderly; repeat dose
MeSH Terms: conditions — Sleep Wake Disorders; Multiple Endocrine Neoplasia Type 1 | interventions — N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: SB-649868 (Experimental): Healthy adult male subjects
  Interventions: Drug: SB-649868
- Cohort 2 (Experimental): Healthy adult female subjects
  Interventions: Drug: SB-649868
- Cohort 3 (Experimental): Healthy male elderly subjects
  Interventions: Drug: SB-649868
- Cohort 4 (Experimental): Healthy female elderly subjects
  Interventions: Drug: SB-649868

INTERVENTIONS:
Drug: SB-649868 — In each of all cohorts, 18 subjects will be randomised in a 2:1 ratio to receive either SB-649868 or placebo

SUMMARY:
The purpose of this study is to determine whether SB-649868 is safe, tolerable after repeated administrations in adult and elderly healthy volunteers. Pharmacokinetics and effects on cardiac function of repeated doses are studied

DETAILED DESCRIPTION:
The present clinical study will assess safety, tolerability and pharmacokinetics of SB-649868 20mg administered for 28 consecutive days in adult (18 to 65 yrs old) and elderly (>65 yrs old) men and women. The study will also assess cardiac function using echocardiography.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. However,

   * Subjects with cTpn I values above 99th percentile of normal range of the selected assay should always be excluded from enrollment;
   * Subjects with AST or ALT > 2xULN should always be excluded from enrollment;
   * Subjects with alkaline phosphatase or bilirubin > 1.5xULN should always be excluded (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
2. Age > or equal to 18 years (applied only to Cohort 1 and 2); age >65 years (applied only to Cohort 3 and 4);
3. Body weight ≥50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive. Slight deviations from these values will be discussed and approved by the Investigator and the GSK Medical Monitor to allow subject inclusion into the study
4. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 3 days post last dose (equivalent to 5 terminal half-lives post-last dose).
5. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their Hormone Replacement Therapy (HRT) during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of contraceptive methods
   * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for 6 weeks following discontinuation of study medication.
6. Having given written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
7. Average QTcB or QTcF < 450 msec; PQ 120-220ms; QRS <120ms; no significant rhythm disorders in SCR 24h Holter-ECG

Exclusion Criteria:

1. History or presence of significant psychiatric, neurological, respiratory, gastrointestinal, hepatic, pancreatic or renal diseases or of any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
2. History of cardiovascular diseases and/or evidence of repolarization defects
3. History of regular alcohol consumption within 6 months of the study defined as:

   • an average weekly intake of greater than 21 units (14 units for female) or an average daily intake of greater than 3 units (2 units for female). 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
4. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
5. Vulnerable subjects , or subject is mentally or legally incapacitated, or language barrier precluding adequate understanding of cooperation.
6. Any history of suicidal behaviour or any suicidal ideation of type 4 or 5 in the last month on the C-SSRS administered at screening
7. Pregnant females as determined by positive Serum beta-hCG test at screening or prior to dosing.
8. Lactating females.
9. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
10. A positive test for HIV antibody.
11. cTpn I values above of 99th percentile of the laboratory reference interval
12. A positive pre-study drug/alcohol screen.
13. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
14. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
15. Consumption of broccoli, radish sprouts, cauliflower, cabbage, orange juice, grapefruit juice or grapefruit within 7 days prior to the first dose of study medication until collection of the final pharmacokinetic blood sample.
16. The subject has participated in a clinical trial and has received an IP within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the IP (whichever is longer).
17. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
18. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
19. Unwillingness or inability to follow the procedures outlined in the protocol.
20. The subject is unable or unwilling to abstain from strenuous physical activity in the 48 h before screening and up to the follow up visit.
21. Subject is the investigator or his/her deputies, research assistant, pharmacist, study coordinator, other staff or relative thereof involved in the conduct of the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-08-27 (Actual); Primary Completion 2010-01-06 (Actual); Study Completion 2010-01-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability evaluated by adverse event monitoring, ECG, vital signs, physical examination, laboratory values (including cTpn I and Insulin) and Romberg/heel to toe test | screening period of 28 days followed by 28 days plus a follow up during 2 weeks approximately

SECONDARY OUTCOMES:
pharmacokinetic after repeat dose. Pharmacodynamic outcomes:Doppler evaluation for tissue velocities, Doppler evaluation of flow, End diastolic and systolic volume and ejection fraction, E/E', and HOMA | within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112861 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112861?search=study&study_ids=112861#rs
- Available data/document: Clinical Study Report: 112861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register